CLINICAL TRIAL: NCT03178890
Title: The Osseointegrated Human-machine Gateway
Brief Title: Osseointegrated Human-Machine Gateway
Acronym: OHMG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Integrum (Industry)
Collaborators: Sahlgrenska University Hospital (Other); Chalmers University of Technology (Other); Vinnova (Other Government); Promobilia Foundation (Other); The Swedish Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 007618
Record Dates: First submitted 2017-02-09; First posted 2017-06-07 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Upper Limb Amputation

STUDY DESIGN:
Intervention Model Description: Prospective study. Each patient is his/her own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osseointegrated Human Machine Gateway (OHMG) (Experimental): Patients will be upgraded to the OHMG if already users of the OPRA Implant System, or implanted with the OPRA Implant System plus OHMG. Each patient will work as his/her own control before and after implantation of the OHMG.
  A single surgery is required to upgrade OPRA Implant System users to the OHMG, and no additional surgeries are required if the OHMG is implanted at the same time as the OPRA Implant System.
  Interventions: Device: OHMG

INTERVENTIONS:
Device: OHMG — Device will be implanted in all enrolled patients.

SUMMARY:
Advanced prosthetic devices are currently controlled by electromyography (EMG) signals generated by patient's stump muscles and recorded by surface electrodes attached on the skin. This way of recordings is often unreliable, inconsistent and leading to high prosthetic abandonment rates for individuals with upper limb amputation. The use of implantable electrodes has been long thought as the solution for a more natural control of artificial limbs, as these offer access to long-term stable and physiologically appropriate sources of control, as well as the possibility to elicit appropriate sensory feedback via neurostimulation.

This Clinical Investigation (CI) is performed to clinically test and verify the safety and benefits of a bidirectional interface into the human body that allows permanent and reliable communication using implanted electrodes. These electrodes will provide long-term stable bioelectric signals for an improved control of artificial limbs. The bidirectional interface is based, and requires, the clinically established implant system for bone-anchored prostheses named Osseointegrated Prostheses for the Rehabilitation of Amputees (OPRA). The feasibility of the device was initially proven through a proof-on-concept patient who has used the system without any adverse events for more than three years.

This CI is performed to verify the safety and benefits of the Osseointegrated Human Machine Gateway (OHMG) as an enhancement of the OPRA Implant System for patients with upper limb amputation, when used within the intended purpose and according to instructions. The CI will be performed at Sahlgrenska University Hospital and Chalmers University of Technology, Sweden. A maximum of eighteen patients will be enrolled. Each patient will undergo a surgery where the OHMG will be implanted. The patients will participate in 8 follow-up sessions, the last one approximately 13 months after the surgery. The study is prospective, where the patient is his/her own control.

ELIGIBILITY:
Inclusion Criteria:

* The patient is an uni- or bi-lateral, transhumeral or transradial amputee
* At least 2 cm from the joint to the most proximal side of the fixture must be present.
* The patient has at least portion of biceps and triceps muscles present.
* The patient currently has, or has been accepted to have, the OPRA Implant System.
* The patient is younger than 70 and older than 17.
* The patient is willing to participate in all assessment sessions (follow-ups).
* The patient has experience using a surface myoelectric prosthesis.

Exclusion Criteria:

* Patient that has a significant cognitive impairment that prevents her/him from following instructions.
* The patient has any concurrent disease or conditions that might affect the treatment with the OHMG.
* The patient is pregnant.
* The patient is participating in another study.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2016-09-26 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of total study population with Adverse Events graded as Serious Adverse Events (SAE) | 13 months
  Serious adverse events are characterized as a) led to death b) led to serious deterioration in health of the subject, that either results in (i) life-threatening illness or injury, (ii) permanent impairment of a body structure or body function, (iii) in-patient or prolonged hospitalization, (iv) medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function or c) led to fetal distress, fetal death or a congenital abnormality or birth defect.
Number of subjects with at least two independent myoelectric signals, and at least one sensory feedback location | 13 months
  For a case to be considered successful in terms of signal transfer; 1) it must be possible to record volitional control of at least two independent muscles with a signal-to-noise ratio of at least 2, and 2) elicit sensory perception via nerve stimulation with a pulse less than 1 milliamperes (mA) amplitude and 1 ms width.
Significant Improvement (p>0,05) in Myoelectric Control Using the "Assessment of Capacity for Myoelectric Control" (ACMC) Functionality Test | 13 months
  All enrolled patients will perform one pre-operative and two post-operative ACMC-tests. The test consists of 30 functional items grouped into 4 hand use areas: gripping, holding, releasing and coordinating. Each person's performance is rated on a 4-pt capability scale. As the items are identified, the rater scores the person's performance on a scale of 0-3 (0 = not capable, 1 = sometimes capable, 2= capable upon request, 3 = spontaneously capable). The results from the pre-operative and post-operative assessments will be statistically analyzed with the Rasch model. Post-operative tests will be conducted 8 and 56 weeks after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Sassu, MD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ortiz-Catalan M, Hakansson B, Branemark R. An osseointegrated human-machine gateway for long-term sensory feedback and motor control of artificial limbs. Sci Transl Med. 2014 Oct 8;6(257):257re6. doi: 10.1126/scitranslmed.3008933. PMID 25298322
- [Background] Branemark R, Berlin O, Hagberg K, Bergh P, Gunterberg B, Rydevik B. A novel osseointegrated percutaneous prosthetic system for the treatment of patients with transfemoral amputation: A prospective study of 51 patients. Bone Joint J. 2014 Jan;96-B(1):106-13. doi: 10.1302/0301-620X.96B1.31905. PMID 24395320